CLINICAL TRIAL: NCT03645096
Title: NCCIH Development of Pregnenolone as a Treatment for Depression R61 Phase
Brief Title: Development of Pregnenolone as a Treatment for Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU 052018-030; 1R61AT009625-01A1 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Pregnenolone; Women
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Pregnenolone; Neurosteroids

STUDY DESIGN:
Intervention Model Description: Adult women with mild to moderate major depressive disorder (MDD) will receive pregnenolone (500 mg/d, 800 mg/d and placebo) in a randomized, double-blind, crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Pregnenolone 500 > Pregnenolone 800 > Placebo (Experimental): 3 exposures in order:
  1. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Matching placebo capsule by mouth, daily for 7 days.
  Interventions: Drug: Pregnenolone 500 mg; Drug: Pregnenolone 800 mg; Drug: Placebo
- Pregnenolone 500 > Placebo > Pregnenolone 800 (Experimental): 3 exposures in order:
  1. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 800 mg capsule by mouth, daily for 7 days.
  Interventions: Drug: Pregnenolone 500 mg; Drug: Pregnenolone 800 mg; Drug: Placebo
- Pregnenolone 800 > Pregnenolone 500 > Placebo (Experimental): 3 exposures in order:
  1. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Matching placebo capsule by mouth, daily for 7 days.
  Interventions: Drug: Pregnenolone 500 mg; Drug: Pregnenolone 800 mg; Drug: Placebo
- Pregnenolone 800 > Placebo > Pregnenolone 500 (Experimental): 3 exposures in order:
  1. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 500 mg capsule by mouth, daily for 7 days.
  Interventions: Drug: Pregnenolone 500 mg; Drug: Pregnenolone 800 mg; Drug: Placebo
- Placebo > Pregnenolone 500 > Pregnenolone 800 (Experimental): 3 exposures in order:
  1. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 800 mg capsule by mouth, daily for 7 days.
  Interventions: Drug: Pregnenolone 500 mg; Drug: Pregnenolone 800 mg; Drug: Placebo
- Placebo > Pregnenolone 800 > Pregnenolone 500 (Experimental): 3 exposures in order:
  1. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 500 mg capsule by mouth, daily for 7 days.
  Interventions: Drug: Pregnenolone 500 mg; Drug: Pregnenolone 800 mg; Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone 500 mg — Pregnenolone 500 mg capsule.
  Other Names: Neurosteroid
Drug: Pregnenolone 800 mg — Pregnenolone 800 mg capsule.
  Other Names: Neurosteroid
Drug: Placebo — Placebo capsule manufactured to mimic pregnenolone capsule.

SUMMARY:
Pregnenolone, an over-the-counter supplement, is a naturally occurring neurosteroid made in the adrenal glands and brain. Preclinical research suggests pregnenolone has antidepressant, cognitive enhancing, and neuroprotective properties, particularly in women. The following hypothesis will be tested in this trial: pregnenolone is associated with improvement in depressive symptom severity in women that is associated with changes in the resting state functional connectivity (rsFC) and GABA.

DETAILED DESCRIPTION:
In this study, 26 adult women meeting criteria for Major Depressive Disorder (MDD) as defined in DSM 5, will be randomized to a double-blind, placebo-controlled, crossover phase I clinical trial of pregnenolone (i.e. each participant receives 500 mg/d, 800 mg/d pregnenolone and placebo in random order). The study will consist of three 7-day treatment exposures to each pregnenolone dose with a 14-day washout between each exposure. Baseline evaluation will include medical and psychiatric history, psychiatric interview, standard laboratory analyses (i.e., blood draw, ECG), and a brief cognitive battery. Neuroimaging will be collected after each study drug or placebo administration. Study drug tolerability and participant safety will be assessed throughout the study (6 in-clinic visits + a safety visit) using structured clinical interviews, self-report questionnaires, and standard laboratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Women, ages 18-65 years, with current MDD (mild or moderate severity per DSM-5) based on SCID-CV.
* No psychotropic medications, other than PRN (as needed) hypnotics, within 28 days of randomization (medication free).
* PRN hypnotics allowed up to 3 days prior to study drug administrations but not while receiving study drug.

Exclusion Criteria:

* Severe MDD based on DSM-5 severity criteria and/or a baseline HRSD score > 27 (consistent with severe depressive symptom severity).
* High risk for suicide (active SI with plan/intent or > 2 lifetime attempts in lifetime or any in the past 6 months).
* Treatment resistant depression (fail two adequate antidepressant trials or ECT during current episode).
* Vulnerable populations (e.g. pregnant/nursing, severe cognitive or intellectual impairment, incarcerated).
* Coronary artery disease, atrial fibrillation, stroke, deep vein thrombosis, pulmonary embolism or blood clotting disorder, or any severe, life threatening or unstable, medical condition.
* History of allergic reaction or side effects with prior pregnenolone use.
* Current substance use disorder defined as meeting criteria for a use disorder based on the SCID interview and self-reported use within the past 3 months, or a positive baseline urine drug screen.
* Current psychotic features (hallucinations, delusions, disorganized thought processes) or eating disorders.
* Anxiety disorders of sufficient severity to be the primary focus of clinical attention (e.g. severe obsessive compulsive or post-traumatic stress disorders).
* Hormone-sensitive conditions (i.e. breast cancer; uterine/ovarian cancer, endometriosis, uterine fibroids).
* Clinically significant laboratory, physical examination, or electrocardiogram (ECG) findings.
* Currently using oral contraceptives containing progestin (barrier methods allowed).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened for eligibility from September 2019 through November 2021 at UT Southwestern in Dallas, TX. 34 Subjects were consented by a research study coordinator in a private office within Dr. Brown's PNE Lab.
Pre-assignment Details: 29 of 34 participants were randomized. It was determined that 5 subjects were not eligible for the study and were not randomized.
Groups:
- Pregnenolone 500 > Pregnenolone 800 > Placebo: 3 exposures in order:
  1. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Matching placebo capsule by mouth, daily for 7 days.
  Pregnenolone 500 mg: Pregnenolone 500 mg capsule.
  Pregnenolone 800 mg: Pregnenolone 800 mg capsule.
  Placebo: Placebo capsule manufactured to mimic pregnenolone capsule.
- Pregnenolone 500 > Placebo > Pregnenolone 800: 3 exposures in order:
  1. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 800 mg capsule by mouth, daily for 7 days.
  Pregnenolone 500 mg: Pregnenolone 500 mg capsule.
  Pregnenolone 800 mg: Pregnenolone 800 mg capsule.
  Placebo: Placebo capsule manufactured to mimic pregnenolone capsule.
- Pregnenolone 800 > Pregnenolone 500 > Placebo: 3 exposures in order:
  1. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Matching placebo capsule by mouth, daily for 7 days.
  Pregnenolone 500 mg: Pregnenolone 500 mg capsule.
  Pregnenolone 800 mg: Pregnenolone 800 mg capsule.
  Placebo: Placebo capsule manufactured to mimic pregnenolone capsule.
- Pregnenolone 800 > Placebo > Pregnenolone 500: 3 exposures in order:
  1. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 500 mg capsule by mouth, daily for 7 days.
  Pregnenolone 500 mg: Pregnenolone 500 mg capsule.
  Pregnenolone 800 mg: Pregnenolone 800 mg capsule.
  Placebo: Placebo capsule manufactured to mimic pregnenolone capsule.
- Placebo > Pregnenolone 500 > Pregnenolone 800: 3 exposures in order:
  1. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 800 mg capsule by mouth, daily for 7 days.
  Pregnenolone 500 mg: Pregnenolone 500 mg capsule.
  Pregnenolone 800 mg: Pregnenolone 800 mg capsule.
  Placebo: Placebo capsule manufactured to mimic pregnenolone capsule.
- Placebo > Pregnenolone 800 > Pregnenolone 500: 3 exposures in order:
  1. Matching placebo capsule by mouth, daily for 7 days followed by 14 day washout.
  2. Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  3. Pregnenolone 500 mg capsule by mouth, daily for 7 days.
  Pregnenolone 500 mg: Pregnenolone 500 mg capsule.
  Pregnenolone 800 mg: Pregnenolone 800 mg capsule.
  Placebo: Placebo capsule manufactured to mimic pregnenolone capsule.
Period: First Treatment (21 Days)
Arm/Group | Pregnenolone 500 > Pregnenolone 800 > Placebo | Pregnenolone 500 > Placebo > Pregnenolone 800 | Pregnenolone 800 > Pregnenolone 500 > Placebo | Pregnenolone 800 > Placebo > Pregnenolone 500 | Placebo > Pregnenolone 500 > Pregnenolone 800 | Placebo > Pregnenolone 800 > Pregnenolone 500
Started | 4 | 4 | 7 | 7 | 5 | 2
Completed | 4 | 3 | 5 | 7 | 3 | 2
Not Completed | 0 | 1 | 2 | 0 | 2 | 0
Period: Second Treatment (21 Days)
Arm/Group | Pregnenolone 500 > Pregnenolone 800 > Placebo | Pregnenolone 500 > Placebo > Pregnenolone 800 | Pregnenolone 800 > Pregnenolone 500 > Placebo | Pregnenolone 800 > Placebo > Pregnenolone 500 | Placebo > Pregnenolone 500 > Pregnenolone 800 | Placebo > Pregnenolone 800 > Pregnenolone 500
Started | 4 | 3 | 5 | 7 | 3 | 2
Completed | 3 | 2 | 5 | 5 | 3 | 2
Not Completed | 1 | 1 | 0 | 2 | 0 | 0
Period: Third Treatment (21 Days)
Arm/Group | Pregnenolone 500 > Pregnenolone 800 > Placebo | Pregnenolone 500 > Placebo > Pregnenolone 800 | Pregnenolone 800 > Pregnenolone 500 > Placebo | Pregnenolone 800 > Placebo > Pregnenolone 500 | Placebo > Pregnenolone 500 > Pregnenolone 800 | Placebo > Pregnenolone 800 > Pregnenolone 500
Started | 3 | 2 | 5 | 5 | 3 | 2
Completed | 3 | 1 | 4 | 3 | 3 | 2
Not Completed | 0 | 1 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants does not differ from the number of participants randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone 500 > Pregnenolone 800 > Placebo | Pregnenolone 500 > Placebo > Pregnenolone 800 | Pregnenolone 800 > Pregnenolone 500 > Placebo | Pregnenolone 800 > Placebo > Pregnenolone 500 | Placebo > Pregnenolone 500 > Pregnenolone 800 | Placebo > Pregnenolone 800 > Pregnenolone 500 | Total
Number analyzed (Participants) | 4 | 4 | 7 | 7 | 5 | 2 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 7 | 7 | 5 | 2 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.50 (7.19) | 43.25 (16.86) | 44.29 (10.94) | 43.71 (11.22) | 46.00 (8.40) | 51.00 (1.41) | 45.62 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 7 | 7 | 5 | 2 | 29
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 3 | 3 | 6 | 6 | 3 | 1 | 22
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 3 | 1 | 1 | 7
  White | 3 | 3 | 5 | 4 | 4 | 1 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 7 | 7 | 5 | 2 | 29
HAM-D [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Rating Scale for Depression (HAM-D) is a 17-item instrument to assess depressive symptom severity. Each item represents a depressive symptom and is scored on a 5-point Likert scale with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = incapacitating. Item scores are summed to derive a total score ranging from 0-68. Higher total scores indicate greater depressive symptom severity.
  units on a scale | 14.75 (2.50) | 12.75 (4.92) | 13.00 (4.28) | 14.14 (5.34) | 16.00 (3.81) | 11.50 (7.78) | 13.90 (4.39)

OUTCOME MEASURES:

1. Primary Outcome: Amygdala-PCC Functional Connectivity
Description: Determine if an increase in Amygdala-PCC functional connectivity is observed with pregnenolone as compared to placebo.
  Amygdala-PCC functional connectivity was measured using resting state fMRI blood-oxygen-level dependent (BOLD) response and transformed to standardized z-scores (with μ=0 and σ=1) for analysis. Functional connectivity was measured three times corresponding to three treatments (500 mg pregnenolone, 800 mg pregnenolone, and placebo). Better outcomes are represented by greater functional connectivity, and are indicated by a higher z-score at 500 mg or 800 mg, relative to that at placebo (i.e., there is no absolute threshold).
Time Frame: 7 days
Population: Some fMRI data may have been unusable due to motion in the scanner.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Pregnenolone (500 mg): Pregnenolone 500 mg capsule by mouth, daily for 7 days.
- Pregnenolone (800 mg): Pregnenolone 800 mg capsule by mouth, daily for 7 days.
- Placebo: Matching placebo capsule by mouth, daily for 7 days.
Arm/Group | Pregnenolone (500 mg) | Pregnenolone (800 mg) | Placebo
Number analyzed (Participants) | 18 | 20 | 18
z-score | -0.0815 (0.1680) | -0.0530 (0.1715) | -0.0456 (0.1736)
Statistical Analysis 1: Comparison: Pregnenolone (500 mg) vs Placebo; Null Hypothesis: Amygdala-PCC functional connectivity (z-score) at 500 mg will be less than or equal to that at placebo. Alternative Hypothesis: Amygdala-PCC functional connectivity (z-score) at 500 mg will be greater than that at placebo; Test type: Superiority; p = .195, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = 0.0493, 95% CI 2-sided [-0.0703 to 0.1689], Standard Error of Mean 0.0554 — Mean Difference = placebo - pregnenolone (500 mg)
Statistical Analysis 2: Comparison: Pregnenolone (800 mg) vs Placebo; Null Hypothesis: Amygdala-PCC functional connectivity (z-score) at 800 mg will be less than or equal to that at placebo. Alternative Hypothesis: Amygdala-PCC functional connectivity (z-score) at 800 mg will be greater than that at placebo; Test type: Superiority; p = .325, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = 0.0262, 95% CI 2-sided [-0.0943 to 0.1467], Standard Error of Mean 0.0565 — Mean Difference = placebo - pregnenolone (800 mg)

2. Primary Outcome: dlPFC-Insula Functional Connectivity
Description: Determine if an increase in dlPFC-Insula functional connectivity is observed with pregnenolone as compared to placebo.
  dlPFC-Insula functional connectivity was measured using resting state fMRI blood-oxygen-level dependent (BOLD) response and transformed to standardized z-scores (with μ=0 and σ=1) for analysis. Functional connectivity was measured three times corresponding to three treatments (500 mg pregnenolone, 800 mg pregnenolone, and placebo). Better outcomes are represented by greater functional connectivity, and are indicated by a higher z-score at 500 mg or 800 mg, relative to that at placebo (i.e., there is no absolute threshold).
Time Frame: 7 days
Population: Some fMRI data may have been unusable due to motion in the scanner.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Pregnenolone (500 mg) | Pregnenolone (800 mg) | Placebo
Number analyzed (Participants) | 18 | 20 | 18
z-score | 0.0495 (0.2524) | 0.1413 (0.3036) | 0.0855 (0.2941)
Statistical Analysis 1: Comparison: Pregnenolone (500 mg) vs Placebo; Null Hypothesis: dlPFC-Insula functional connectivity (z-score) at 500 mg will be less than or equal to that at placebo. Alternative Hypothesis: dlPFC-Insula functional connectivity (z-score) at 500 mg will be greater than that at placebo; Test type: Superiority; p = .468, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = -0.0071, 95% CI 2-sided [-0.1969 to 0.1827], Standard Error of Mean 0.0878 — Mean Difference = placebo - pregnenolone (500 mg)
Statistical Analysis 2: Comparison: Pregnenolone (800 mg) vs Placebo; Null Hypothesis: dlPFC-Insula functional connectivity (z-score) at 800 mg will be less than or equal to that at placebo. Alternative Hypothesis: dlPFC-Insula functional connectivity (z-score) at 800 mg will be greater than that at placebo; Test type: Superiority; p = .458, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = 0.0097, 95% CI 2-sided [-0.1803 to 0.1996], Standard Error of Mean 0.0891 — Mean Difference = placebo - pregnenolone (800 mg)

3. Primary Outcome: GABA Concentration.
Description: Determine if an increase in occipital GABA concentration is observed with pregnenolone, as compared to placebo.
  Occipital GABA concentration using spectroscopy with tCr reference. Higher concentration values are representative of a greater anti-depressant effect.
Time Frame: 7 days
Population: All participants with available data for each treatment condition.
Measure: Mean (Standard Deviation); unit: millimolars (mM)
Arm/Group | Pregnenolone (500 mg) | Pregnenolone (800 mg) | Placebo
Number analyzed (Participants) | 17 | 19 | 18
millimolars (mM) | 0.0947 (0.0294) | 0.0861 (0.0264) | 0.0974 (0.0262)
Statistical Analysis 1: Comparison: Pregnenolone (500 mg) vs Placebo; Null Hypothesis: GABA concentration (mM) at 500 mg will be less than or equal to that at placebo. Alternative Hypothesis: GABA concentration (mM) at 500 mg will be greater than that at placebo; Test type: Superiority; p = .316, t-test, 1 sided — Paired samples t-test with corrected standard deviation of the difference; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = 0.0038, 95% CI 2-sided [-0.0132 to 0.0209], Standard Error of Mean 0.0078 — Mean Difference = placebo - pregnenolone (500 mg)
Statistical Analysis 2: Comparison: Pregnenolone (800 mg) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .071, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = 0.0131, 95% CI 2-sided [-0.0050 to 0.0312], Standard Error of Mean 0.0084 — Mean Difference = placebo - pregnenolone (800 mg)

4. Secondary Outcome: Pregnenolone Level
Description: Assess bioavailability of pregnenolone by demonstrating increases in serum pregnenolone and allopregnanolone with pregnenolone administration. Change (increases) in blood serum pregnenolone levels are indicative of bioavailability.
Time Frame: 7 days
Population: All participants with available data for each treatment condition.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Placebo: Matching placebo capsule by mouth, daily for 7 days.
  .
Arm/Group | Pregnenolone (500 mg) | Pregnenolone (800 mg) | Placebo
Number analyzed (Participants) | 16 | 19 | 17
pg/mL | 10902.60 (11849.18) | 11484.75 (13038.50) | 769.63 (554.50)
Statistical Analysis 1: Comparison: Pregnenolone (500 mg) vs Placebo; Null Hypothesis: Pregnenolone level (pg/mL) at 500 mg will be less than or equal to that at placebo. Alternative Hypothesis: Pregnenolone level (pg/mL) at 500 mg will be greater than that at placebo; Test type: Superiority; p = .006, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = -11322.45, 95% CI 2-sided [-19577.27 to -3067.62], Standard Error of Mean 3750.52 — Mean Difference = placebo - pregnenolone (500 mg)
Statistical Analysis 2: Comparison: Pregnenolone (800 mg) vs Placebo; Null Hypothesis: Pregnenolone level (pg/mL) at 800 mg will be less than or equal to that at placebo. Alternative Hypothesis: Pregnenolone level (pg/mL) at 800 mg will be greater than that at placebo; Test type: Superiority; p = .003, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = -11828.78, 95% CI 2-sided [-19650.24 to -4007.33], Standard Error of Mean 3620.42 — Mean Difference = placebo - pregnenolone (800 mg)

5. Secondary Outcome: Allopregnanolone Level
Description: Assess bioavailability of pregnenolone by demonstrating increases in serum pregnenolone and allopregnanolone with pregnenolone administration. Change (increases) in blood serum allopregnanolone levels are indicative of bioavailability.
Time Frame: 7 days
Population: All participants with available data for each treatment condition.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pregnenolone (500 mg) | Pregnenolone (800 mg) | Placebo
Number analyzed (Participants) | 16 | 19 | 17
pg/mL | 2478.39 (1801.67) | 2489.08 (2180.59) | 124.22 (224.62)
Statistical Analysis 1: Comparison: Pregnenolone (500 mg) vs Placebo; Null Hypothesis: Allopregnanolone level (pg/mL) at 500 mg will be less than or equal to that at placebo. Alternative Hypothesis: Allopregnanolone level (pg/mL) at 500 mg will be greater than that at placebo; Test type: Superiority; p = .001, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = -2523.58, 95% CI 2-sided [-3724.93 to -1322.22], Standard Error of Mean 545.83 — Mean Difference = placebo - pregnenolone (500 mg)
Statistical Analysis 2: Comparison: Pregnenolone (800 mg) vs Placebo; Null Hypothesis: Allopregnanolone level (pg/mL) at 800 mg will be less than or equal to that at placebo. Alternative Hypothesis: Allopregnanolone level (pg/mL) at 800 mg will be greater than that at placebo; Test type: Superiority; p = .001, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = -2480.62, 95% CI 2-sided [-3739.32 to -1221.93], Standard Error of Mean 582.63 — Mean Difference = placebo - pregnenolone (800 mg)

6. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE)
Description: Assess safety and tolerability of pregnenolone at the doses tested.
  SAFTEE is a side effect self-report assessment scale that consists of 56 potential side effects. Participants rate how bothersome each side effect is on a scale of "none" (0), "mild" (1), "moderate" (2), "severe" (3). Total scores range from 0 to 168. A higher total score (sum of all items) indicates a higher level of side effect burden.
Time Frame: 7 days
Population: All participants with available data for each treatment condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone (500 mg) | Pregnenolone (800 mg) | Placebo
Number analyzed (Participants) | 20 | 22 | 20
units on a scale | 16.15 (12.42) | 19.14 (12.41) | 17.60 (9.65)
Statistical Analysis 1: Comparison: Pregnenolone (500 mg) vs Placebo; Null Hypothesis: SAFTEE (total) scores at 500 mg will be greater than or equal to that at placebo. Alternative Hypothesis: SAFTEE (total) scores at 500 mg will be less than that at placebo; Test type: Non-Inferiority — Using the two one-sided test (TOST) procedure (Schuirmann, 1987), equivalence is established at the α significance level if a (1-2α) × 100% confidence interval for the difference in efficacies (new - current) is contained within the interval (-δ, δ) Schuirmann, D. J. (1987). A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. Journal of pharmacokinetics and biopharmaceutics, 15, 657-680; p = .336, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = 0.7059, 95% CI 2-sided [-2.7659 to 4.1777], Standard Error of Mean 1.6377 — Mean Difference = placebo - pregnenolone (500 mg)
Statistical Analysis 2: Comparison: Pregnenolone (800 mg) vs Placebo; Null Hypothesis: SAFTEE (total) scores at 800 mg will be greater than or equal to that at placebo. Alternative Hypothesis: SAFTEE (total) scores at 800 mg will be less than that at placebo; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = .240, t-test, 1 sided — Statistical significance is evaluated at p (one-tailed) <= .05; Paired samples t-test with corrected standard deviation of the difference; Mean Difference (Final Values) = -2.5000, 95% CI 2-sided [-9.8131 to 4.8131], Standard Error of Mean 3.4662 — Mean Difference = placebo - pregnenolone (800 mg)

7. Secondary Outcome: Pregnenolone Dose
Description: Identify a dose of pregnenolone that demonstrates bioavailability (see "Pregnenolone Level" and "Allopregnanolone Level" outcome measures), tolerability (see "SAFTEE" outcome measure); and is associated with a significant change in a biosignature.
Time Frame: 7 days
Measure: Number; unit: mg
Groups:
- Pregnenolone Arm: This arm includes all participants who received the different doses of the intervention (i.e., Pregnenolone 500mg and 800 mg, *not* including placebo)
  Pregnenolone 500 mg capsule by mouth, daily for 7 days.
  Pregnenolone 800 mg capsule by mouth, daily for 7 days.
Arm/Group | Pregnenolone Arm
Number analyzed (Participants) | 21
mg | 500

ADVERSE EVENTS:
Time Frame: AEs were collected over a 2+ year period.
Groups:
- Pregnenolone 800: Pregnenolone 800 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  Pregnenolone 800 mg: Pregnenolone 800 mg capsule.
- Pregnenolone 500: Pregnenolone 500 mg capsule by mouth, daily for 7 days followed by 14 day washout.
  Pregnenolone 500 mg: Pregnenolone 500 mg capsule.
Arm/Group | Pregnenolone 800 | Pregnenolone 500 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
Some fMRI data may have been excluded as a result of motion in the MRI machine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT03645096/Prot_SAP_000.pdf